CLINICAL TRIAL: NCT06660082
Title: Early Rehabilitation Using Head Impulse Test for Acute Vestibular Deficit
Acronym: KINE HIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL24_0718; 2024-A02268-39 (Other: ID-RCB)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Vestibular Schwannoma; Unilateral Vestibular Deficit
Keywords: Vestibular rehabilitation; Vestibular schwannoma; Vestibulo-ocular Reflex (VOR); video Head Impulse Test (vHIT)
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Head Movements

STUDY DESIGN:
Intervention Model Description: Exploratory, single-centre, randomised, sham-controlled, single-blind, superiority study, with comparison of two groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be aware of the experimental or sham status of the arm they'll be allocated to.
  Investigator realising offline analysis will not know the arm of allocation of the subject they are analysing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants included in this group will undergo experimental treatment as described below.
  Head movements
  Interventions: Procedure: Experimental treatment: Head movements
- Control Group (Sham Comparator): Participants included in this group will undergo sham-treatment as described below.
  Eye movements without head movements
  Interventions: Procedure: Sham treatment: only eye movements

INTERVENTIONS:
Procedure: Experimental treatment: Head movements — These are gaze stabilisation exercises under vHIT control, between post-operative days 1 to 6.
  The patient sits facing a wall 2 metres away. The investigator places the vHIT device on the participant's head and ensures that it fits properly.
  This is followed by an initial calibration phase (the patient must follow a laser dot with his eyes).
  Then comes stimulation phase: the investigator, standing behind the patient, places his hands on the sides of the patient's lower jaw, which he is asked to clench. The investigator asks the subject to stare at a visual target on the wall in front of the patient. The investigator then performs a series of low-amplitude, high-speed head movements in the plane of the lateral canals and on the side of the vestibular deficit.
  The patient is encouraged to resume fixation of the visual target as quickly as possible.
  For each treatment session, patients should perform a minimum of 10 impulses and a maximum of 30 impulses on the deafferented side. Each
  Other Names: Head movements
  Arms: Experimental Group
Procedure: Sham treatment: only eye movements — These are visually guided saccade exercises under vHIT device control but without head movements (saccade module), between post-operative days 1 to 6.
  For this sham treatment, the modalities are identical to the experimental treatment session, up to the calibration phase described above.
  For the stimulation phase, the investigator, standing behind the patient, places his hands on the sides of the patient's lower jaw, which he is asked to clench. The investigator asks the subject to stare at a visual target on the wall in front of the patient. The target then jumps horizontally to trigger visually guided saccades or slides horizontally to trigger an eye-tracking movement. The investigator stabilises the patient's head to prevent any head movement. The patient is encouraged to resume or maintain fixation of the visual target as quickly as possible.
  A minimum of 5 horizontal saccade sequences and 5 horizontal eye-tracking sequences will be performed. Each training session lasts approxi
  Arms: Control Group

SUMMARY:
The vestibulo-ocular reflex (VOR) induces a compensatory movement in the eye when the head is rotated, to maintain stable vision when we move. It originates in the peripheral vestibular system, which detects head movements. It is particularly effective for rapid head movements, as tested in the Head Impulse Test (HIT). In acute unilateral vestibular deficit (AUVD), the VOR deficit is compensated for by a substitution saccade, more commonly known as catch up saccade, that contribute to refocus the gaze and maintain vision during head rotations.

Recent technological advances have made it possible to make high-quality recordings during HIT (video Head Impulse Test, vHIT), leading to the identification of substitution saccades of variable latency. Our team has shown that saccades of shorter latency lead to better visual function (Hermann et al., 2017) and that the cerebellum is involved in the development of these saccades (Hermann et al., 2023), suggesting a learning effect rather than the de novo appearance of particular saccades.

The main hypothesis of this study is that the mechanisms underlying short-latency substitution saccades, which seems to guarantee good functional recovery, depend on learning occurring from the first days after an acute unilateral vestibular deficit. We also hypothesise that early physiotherapeutic rehabilitation of the VOR under Head Impulse Test conditions would promote this learning process and the development of early catch-up saccades.

One of the causes of AVD is the resection of cochleovestibular schwannomas. This procedure involves a neurotomy, i.e. complete vestibular deafferentation, which is precisely known due to the scheduled nature of the surgery. The exact moment of onset of vestibular damage is therefore known, unlike other vestibular pathologies. Hospitalisation is necessary in the immediate aftermath of surgery, with the presence of physiotherapists on the wards. In addition, there is no spontaneous recovery of the vestibular deficit. These patients therefore represent the ideal acute unilateral vestibular deficit model for testing our hypothesis. Two studies using vHIT in the aftermath of vestibular schwannoma resection surgery (Pogson et al. 2022; Mantokoudis et al. 2014) also allow us to confirm the safety and feasibility of our protocol in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral vestibular schwannoma and programmed surgery
* vestibulo-ocular reflex gain :

  * on pathological side > 0.50
  * on healthy side > 0.80
* all information's concerning the study given more than 15 days before surgery and consent collected the day before surgery

Exclusion Criteria:

* Radiotherapy treatment prior to surgery.
* Resumption of surgery
* Presence of bilateral vestibular schwannomas
* Normal or Corrected to normal distance visual acuity < 5/10
* Presence of other aetiologies that may explain the ataxic syndrome and/or oscillopsias
* Oculomotor paralysis, ocular instability in primary position
* Use of medications that compromise eye movement (psychotropic drugs)
* Cervical spinal pathology with instability (contraindication for vHIT)
* Cochlear implantation
* Non-stabilized medical condition
* Pregnant women. This exclusion criterion will be investigated by questioning the patient.
* Patient under guardianship
* Patient not affiliated to a social security scheme
* Patient participating any other interventional study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
First Substitution Saccade Latency after treatment | Day 7
  Mean latencies (in milliseconds) of the first substitution saccade assessed by vHIT examination, in both groups.
  Eye movements are recorded during the vHIT examination, carried out by one of the expert practitioners (physiotherapist or doctor) investigating the study. Data from the vHIT are extracted, enabling offline analysis of oculomotor parameters, including the latency of the first substitution saccade in milliseconds. These analyses are carried out off-line by the principal investigator, who was trained and experienced in this type of analysis, using software that allowed standardised and automated analysis, blinded to the group.

SECONDARY OUTCOMES:
First Substitution Saccade Latency during the First Week | Everyday from post-surgery Day 1 to Day 6
  Mean latencies (in milliseconds) of the first substitution saccade assessed by vHIT examination, in the experimental group.
  This secondary outcome measure is analysed using the same method described for Main Outcome
First Saccade Latency after treatment (follow-up) | At post-surgery Day 45 and 3rd month
  Mean latencies (in milliseconds) of the first substitution saccade assessed by vHIT examination, for both groups
  This secondary outcome measure is analysed using the same method described for Main Outcome
First saccades amplitude after treatment | Post surgery Day 7, Day 45 and 3rd month
  Mean amplitudes (degrees) of the first substitution saccade assessed by vHIT examination, in both groups.
  Eye movements are recorded during the vHIT examination, carried out by one of the expert practitioners (physiotherapist or doctor) investigating the study. Data from the vHIT are extracted, enabling offline analysis of oculomotor parameters, including the amplitude of the first substitution saccade in milliseconds. These analyses are carried out off-line by the principal investigator, who was trained and experienced in this type of analysis, using software that allowed standardised and automated analysis, blinded to the group.
First saccades amplitude during first week | Everyday from post-surgery Day 1 to Day 6
  Mean amplitudes (degrees) of the first substitution saccade assessed by vHIT examination, in the experimental group
  This secondary outcome measure is analysed using the same method described for Main Outcome.
Balance and gait assessment | At Day -1 (pre-surgery), and post-surgery Day 7, Day 45 and 3rd Month
  Score of the modified Dynamic Gait index (m-DGI), in both groups.
Quality of Life Assessment | At Day -1 (pre-surgery), and post-surgery Day 7, Day 45 and 3rd Month
  Score of the self administered Dizziness handicap Inventory (DHI), in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Pierre Wertheimer Hospital - Neurological Hospital, Bron, France

IPD SHARING:
Plan to Share IPD: No